CLINICAL TRIAL: NCT05334953
Title: Comparing the Efficacy of Extracorporeal Shock Wave Therapy, Ultrasound and Phonophoresis Treatments in Lateral Epicondylitis: A Randomized Controlled Trial
Brief Title: Efficacy of Extracorporeal Shock Wave Therapy, Ultrasound and Phonophoresis Treatments in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 71306642-050.05.04
Record Dates: First submitted 2022-03-31; First posted 2022-04-19 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis; extracorporeal shock wave therapy; ultrasound; phonophoresis
MeSH Terms: conditions — Tennis Elbow | interventions — Phonophoresis; Ultrasonography; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: ESWT(Extracorporeal Shock Wave Therapy) (Experimental): Group 1 (n = 17) will be given two times a week, total 5 sessions of ESWT + home exercise program
  Interventions: Device: ESWT
- Phonophoresis (Experimental): Group 2 ( n=17) will be given five times a week, total 10 sessions of diclofenac phonophoresis + home exercise program
  Interventions: Device: Phonophoresis
- Ultrasound therapy (Experimental): Group 2 (n=17) will be given five times a week, total 10 sessions of ultrasound therapy+ home exercise program
  Interventions: Device: Ultrasound
- Control goup (Other): Group 4 ( n=17) will be given home exercise program
  Interventions: Other: Control group

INTERVENTIONS:
Device: ESWT — Group 1 (n = 17) will be given two times a week, total 5 sessions of ESWT + home exercise program
  Other: Home Workout Program Patients will be given eccentric exercises and stretching exercises
  Arms: Experimental: ESWT(Extracorporeal Shock Wave Therapy)
Device: Phonophoresis — Group 2 ( n=17) will be given five times a week total 10 sessions of diclofenac phonophoresis + home exercise program
  Other: Home Workout Program Patients will be given eccentric exercises and stretching exercises
  Arms: Phonophoresis
Device: Ultrasound — Group 3 (n=17) will be given five times a week total 10 sessions of ultrasound therapy+ home exercise program
  Other: Home Workout Program Patients will be given eccentric exercises and stretching exercises
  Arms: Ultrasound therapy
Other: Control group — Other: Home Workout Program Patients will be given eccentric exercises and stretching exercises
  Arms: Control goup

SUMMARY:
The aim of this study; to determine the effectiveness of ESWT, ultrasound and phonophoresis treatments on pain, grip strength, functionality and quality of life in patients with lateral epicondylitis and to determine the superiority of the treatments to each other.

DETAILED DESCRIPTION:
Lateral epicondylitis is the most common cause of elbow lateral pain in adults. Pain that occurs in LE and radiates to the humerus and forearm is characteristic of this disease. The main complaints being pain and decreased grip strength, both of which may affect activities of daily living. The patient's complaints regress with rest,but but can increase again during daily activities such as grasping, repetitive hand movements, holding door handles, turning keys, lifting heavy loads. Diagnosis of lateral epicondylitis is largely based on clinical history and examination. Conservative treatment is the first line treatment. Generally, %90 of patients with LE benefit from conservative and medical treatment, and only a few need surgery. These treatment methods include many options such as activity modification, topical and oral NSAIDs, splinting, stretching and strengthening exercises, various injections, prolotherapy and electrotherapy modalities. Laser, TENS, ultrasound, phonophoresis, iontophoresis and ESWT are electrotherapeutic agents that can be used in therapy to relieve pain and promote healing. Research on physical treatments for LE has not yet proven superiority of one specific approach.

Although many studies have been done for ESWT, ultrasound and phonophoresis, there is not any study that compares these three modalities.In addition, there ara fewer studies about measuring the effect of these treatment methods which contain control groups. In this study, our aim is to investigate the efficacy of ESWT, ultrasound therapy and phonophoresis methods used in the treatment of LE and to compare the efficacy of these three treatments against each other and control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years
* Pain on the lateral side of the elbow for at least 4 weeks
* Tenderness over the lateral epicondyle
* Positive in at least two of the lateral epicondylitis spesific tests (Cozen test, Maudley test and Mills test)

Exclusion Criteria:

* Be younger than 18
* Having had ESWT treatment in the elbow area before
* History of injection, surgery, physical therapy in the elbow area in the last 3 months
* Previous elbow surgery
* History of radius/ulna fracture
* A history of cervical and shoulder problems
* having bilateral symptoms
* concomitant medial epicondylitis
* Malignancy
* Pregnancy
* Systemic rheumatologic disease or systemic infection
* inserted cardiac pacemaker
* presence of coagulation disorders
* Cognitive disfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Change from Baseline at 1 month after treatment.
  The self-evaluation of pain severity during rest, activity,night and with palpation was calculated using a 10-cm VAS scale

SECONDARY OUTCOMES:
Patient-Rated Tennis Elbow Evaluation (PRTEE) scales | Change from Baseline at 1 month after treatment.
  The PRTEE is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire score | Change from Baseline at 1 month after treatment.
  The Quick DASH is an 11-item measure of the magnitude of disability and symptoms specific to the upper extremity. The first 6 items measure the degree of difficulty in performing various physical activities because of a shoulder, arm, and hand problem, and the other 5 items related to quality of sleeping, social activities, and daily activities, and the intensity of pain and numbness
Roles and Maudsley Score | Change from Baseline at 1 month after treatment.
  The Roles and Maudsley score was used to evaluate pain and activity limitation as classified in four categories: 1 point = excellent, 2 points = good, 3 points = fair and 4 points = poor.
Health Assessment Questionnaire (HAQ) score | Change from Baseline at 1 month after treatment.
  This is a self-reported questionnaire covering 20 items in eight domains related to measuring difficulty in performing activities of daily living: dressing, arising, eating, walking, hygiene, reach, grip, and common daily activities
Grip Strength score | Change from Baseline at 1 month after treatment.
  Grip strength of the affected upper extremity was calculated using a Hydraulic Hand Dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Okan Küçükakkaş, Doç, Study Director — okan4494@yahoo.com; Elif Uğurlu, MD, Principal Investigator — elifdemirbag92qgmail.com
Locations (1):
- Bezmialem Vakif university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yalvac B, Mesci N, Geler Kulcu D, Yurdakul OV. Comparison of ultrasound and extracorporeal shock wave therapy in lateral epicondylosis. Acta Orthop Traumatol Turc. 2018 Sep;52(5):357-362. doi: 10.1016/j.aott.2018.06.004. Epub 2018 Jun 28. PMID 30497658
- [Background] Bayram K, Yesil H, Dogan E. Efficacy of extracorporeal shock wave therapy in the treatment of lateral epicondylitis. North Clin Istanb. 2014 Aug 3;1(1):33-38. doi: 10.14744/nci.2014.77487. eCollection 2014. PMID 28058299
- [Background] Stasinopoulos D, Johnson MI. Cyriax physiotherapy for tennis elbow/lateral epicondylitis. Br J Sports Med. 2004 Dec;38(6):675-7. doi: 10.1136/bjsm.2004.013573. PMID 15562158
- [Background] Weber C, Thai V, Neuheuser K, Groover K, Christ O. Efficacy of physical therapy for the treatment of lateral epicondylitis: a meta-analysis. BMC Musculoskelet Disord. 2015 Aug 25;16:223. doi: 10.1186/s12891-015-0665-4. PMID 26303397